CLINICAL TRIAL: NCT06220084
Title: Therapeutic Dance in Parkinson's Disease: The UPbeating GReek Application of DancE in Parkinson's Disease (UPGRADE-PD) Clinical Trial
Brief Title: The UPbeating GReek Application of DancE in Parkinson's Disease Clinical Trial
Acronym: UPGRADE-PD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of West Attica (Other)
Collaborators: World in Harmony/Mundo en Armonia (Unknown)
Responsible Party: Principal Investigator, Michail Elpidoforou, Principal Investigator, University of West Attica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 92282/10.10.2023; 688/07.09.2022 (Registry Identifier: Eginition's Hospital Ethics Committee)
Record Dates: First submitted 2023-12-29; First posted 2024-01-23 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Dance; Dance for Parkinson's; Quality of Life; Depression; Fatigue; Cognitive Functions; Stress; Anxiety; Frailty; Sarcopenia; Body Mass Index; Balance; Music Preferences
MeSH Terms: conditions — Parkinson Disease; Depression; Fatigue; Anxiety Disorders; Frailty; Sarcopenia

STUDY DESIGN:
Intervention Model Description: Groups: live DfPD® vs remote DfPD® vs Control. The experimental period will be of 10 months, including 3 periods of two months intervention for each group (live DfPD® vs remote DfPD®) versus control group (non-intervention group) and 2 washout periods of two months between.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Live DfPD® (Experimental): Eight weeks intervention of two 60min live dance classes per week plus their usual care
  Interventions: Behavioral: Dance for PD®
- Remote DfPD® (Experimental): Eight weeks intervention of two 60min online-via zoom platform dance classes per week plus their usual care
  Interventions: Behavioral: Dance for PD®
- Control (No Intervention): Non-interventional group in which participants receive their usual care only

INTERVENTIONS:
Behavioral: Dance for PD® — The intervention consists of 16 60-min adapted to Greek culture DfPD® classes, which will be performed twice weekly for 8 weeks and instructed by a single researcher, who has the approval to use it for research reasons. The intervention will be delivered both live and online in separate periods for each participant.
  Other Names: Dance for Parkinson's®, DfPD®
  Arms: Live DfPD®; Remote DfPD®

SUMMARY:
Dance for Parkinson's Disease® (DfPD®) is a specially designed dance program for individuals with PD. This study assesses the efficacy, safety and feasibility of a culturally adapted DfPD® program offered both live and online in Greek PD patients.

A total of 40 early-to-mid-stage PD Greek patients have been enrolled to underwent a total of 16 60-min classes twice weekly over 8 weeks both live and online as well as to be part of the non-intervention control group in a 3-arms crossover randomized controlled clinical trial. Assessments will be performed at baseline and at the end of each study period and will include quality of life, fatigue, depressive symptoms, stress, anxiety, sarcopenia, frailty, balance, cognitive functions, movement and non-movement PD symptoms, and Body Mass Index (BMI). Safety and feasibility of each of the dance interventions (live DfPD® vs remote DfPD®) will be assessed.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is an idiopathic, neurodegenerative, and progressive movement disorder in which several types of physical exercise seem to have positive effects. Dance, as a form of organized physical activity, seems to more easily motivate PD patients to attend exercise classes with higher compliance rates and lower dropout rates in comparison with other means of exercise.

Dance for Parkinson's Disease® (DfPD®, or Dance for PD®) is a structured therapeutic dance program for people with PD designed by the Brooklyn Parkinson Group (BPG) and the Mark Morris Dance Group (MMDG) in 2001. The positive effect of the above program has been already shown for several factors, such as Quality of Life (QoL), motor functions, cognition, self-efficacy, anxiety, depression, and fatigue in PD patients. To our knowledge, there is no study investigating the effect of DfPD® on PD patients' frailty and sarcopenia. In addition, no randomized controlled clinical study to date has been conducted to investigate the effect of DfPD® on Greek PD patients to any parameter.

The main research purpose of that study is to investigate the possible positive effects of DfPD® in QoL, fatigue, depressive symptoms, stress, anxiety, sarcopenia, frailty, balance, cognitive functions, movement and non-movement PD symptoms, and Body Mass Index (BMI) of Greek Parkinson's individuals. The above scientific study is a 3-arms crossover randomized controlled clinical trial (live DfPD® vs remote DfPD® vs Control), and the experimental period will be of 10 months, including 3 periods of two months intervention of two 60min dance classes per week for each group (live DfPD® vs remote DfPD®) versus control group (non-intervention group) and 2 washout periods of two months between.

A total of 40 early-to-mid-stage PD Greek patients have been enrolled to underwent a total of 16 60-min classes twice weekly over 8 weeks both live and online as well as to be part of the non-intervention control group. Assessments will be performed at the baseline and at the end of each period (6 in total per individual) for each of the above parameters. Safety and feasibility will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* An established diagnosis of idiopathic PD of an early-to-moderate severity; that is from 0 to 2,5 according to Hoehn and Yahr (H&Y) stages
* Ability to understand, write, and speak in Greek
* Written consent for participating into the study
* Smart device (either smart phone or tablet/laptop/computer) access for the dance intervention which will be conducted remotely

Exclusion Criteria:

* A diagnosis of a non-PD tremor disorder
* Moderate-to-severe PD (≥3 H&Y stages), due to a high falls risk
* Serious health or disability issues (either physical or mental), due of which exercise is not permitted and/or basic instructions during the program cannot be followed
* Mental disorder not related to PD
* Any disease other than PD, which could affect mobility levels
* Any electronic internal medical device or implant, such as a pacemaker or a deep brain stimulation, due to contraindication in the use of bio-electrical impedance analysis
* No access of the participant or patient's carer to any smart device (either smart phone or tablet/laptop/computer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2024-07-11 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in total score of Parkinson's Disease Questionnaire-8 (PDQ-8) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Minimum score 0, Maximum score 100. A higher score indicates worse quality of life.

SECONDARY OUTCOMES:
Change in total score of Parkinson Fatigue Scale-16 (PFS-16) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Minimum score 1, Maximum score 5. A higher score indicates more fatigue.
Change in total score of Modified Fatigue Impact Scale (MFIS) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Minimum score 0, Maximum score 84. A higher score indicates more fatigue.
Change in total score of Montreal Cognitive Assessment (MoCA) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Minimum score 0, Maximum score 30. Lower scores indicate cognitive impairment.
Change in total score of Berg Balance Scale (BBS) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Minimum score 0, Maximum score 56. Lower scores indicate worse balance.
Change in Depression Score of Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Normal score 0-9, Mild score: 10-12, Moderate score: 13-20, Severe score: 21-27, and Extremely severe: 28-42
Change in Anxiety Score of Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Normal score 0-6, Mild score: 7-9, Moderate score: 10-14, Severe score: 15-19, and Extremely severe: 20-42
Change in Stress Score of Depression, Anxiety and Stress Scale 21 (DASS-21) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  Normal score 0-10, Mild score: 11-18, Moderate score: 19-26, Severe score: 27-34, and Extremely severe: 35-42
Change in Patient Outcomes using the Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  MDS-UPDRS has 4 parts. Part I assesses non-motor experiences of daily living (13 items, score range: 0-52), part II assesses motor experiences of daily living (13 items, score range: 0-52), part III assesses motor signs (33 items, score range: 0-132), and part IV assesses motor complications, dyskinesias and motor fluctuations (6 items, score range: 0-24). Each item score ranges from 0 (normal) to 4 (severe) and higher scores indicate a greater impact of Parkinson's disease signs.
Change in total score of SARC-F Scale | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  SARC-F is a self-reporting screening tool for the assess of the sarcopenia risk and comprises five components: strength, assistance walking, rise from a chair, climb stairs, and number of falls (score range: 0-2 for each component, and 0-10 in total. Healthy status score range: 0-3, risk of sarcopenia score: ≥4).
Change in Sarcopenia status using the European Working Group on Sarcopenia in Older People (EWGSOP2) criteria | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  According to EWGSOP2, sarcopenia is (a) probable to an individual with low muscle strength (hand grip strength for men: <27 kg, and women: <16 kg), (b) confirmed to an individual with the above criteria plus low muscle quantity (appendicular skeletal muscle mass index for men: <7 kg/m^2, and women: <5,5 kg/m^2), and (c) severe to an individual with the two above criteria plus low physical performance (4-m usual walking speed test ≤0.8 m/s). Hand grip strength will be assessed by a calibrated digital handheld dynamometer, appendicular muscle mass index by a bioelectrical impedance analysis (BIA) equipment, and physical performance by the 4-min usual walking speed test.
Change in Body Mass Index | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  A score from the equation kg/m^2. Lower scores than 18,5 indicate underweight, scores of 18,5-24,9 indicate normal weight, scores of 25-29,9 indicate overweight and scores equal or over 30 indicate obesity. Within the obesity category 3 subcategories exist: Class I scores of 30-34, Class II scores of 35-39, and Class III scores of ≥40.
Changes in Frailty Phenotype (FP) status | Baseline, 10 weeks, 19 weeks, 28 weeks, 37 weeks, and 46 weeks.
  According to the Fried FP, 5 criteria have to be assessed: unintentional weight loss >5 kg the last year, weakness (handgrip strength for men: <27 kg, and women: <16 kg), slow walking speed (10-m usual walking speed test ≤0.8 m/s), exhaustion (PFS-16 total score ≥3, which indicates moderate-to-severe fatigue), and low levels of physical activity (International Physical Activity Questionnaire-Short Form/IPAQ-SF total score <600 MET-min-week^-1, which indicates inactivity). The FP score ranges from 0 to 5 (1 point for each criteria; 0: best score to 5: worst score). As frail defined an individual with a score of ≥3, as pre-frail an individual with a score of 1-2, and as non-frail or robust an individual with a score 0.
Registration of Music Preferences via Music Preferences Scale of Gardikiotis & Baltzis | Baseline (week 1)
  Music Preferences scale of Gardikiotis & Baltzis is a 6-point Likert scale (0: i don't know it, 1: i don't like it at all to 5: i like it very much) of 24 items (each item includes a different music genre) and evaluates the individual's level of preference to a variety of Greek and non-Greek music.

OTHER OUTCOMES:
Occurence of Adverse Events and Emergent Adverse Events | During the interventional periods (live DfPD® and remote DfPD®) for each participant.
  Occurence of adverse events comprising falls, injuries, muscle soreness or excessive fatigue, and emergent adverse events comprising death, life-threatening, hospitalization, persistent or significant disability, congenital anomaly/birth defect or necessity of surgical operation for any of the above.
Adherence and Attrition Assessment | During the intervention (week 2-45)
  Adherence and attrition rates; an adherence rate ≥70% is considered as high in elderly with functional limitations, and attrition rate ≤15% is considered acceptable by the PEDro scale.
Assessment of Patient's Satisfaction | End of the program (week 45)
  Verbal statement for willingness to continue the program after the end of the intervention in a 6-point Likert scale (0: i don't know if i'd like to continue the program, 1: i don't want to continue the program at all to 5: i want to continue the program very much), and two open questions (I. Could you please list all the positive and negative points of the live DfPD® intervention? and II. Could you please list all the positive and negative points of the online DfPD® intervention?) in a 1-to-1 interview for each participant in the end of the program.
Assessment of Recruitment Rates | Start of Recruitment (-6 months), Baseline (week 1)
  Target, up to 5 months for 40 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Michail Elpidoforou, MSc, Principal Investigator — Laboratory of Neuromuscular and Cardiovascular Study of Motion (LANECASM)
Locations (1):
- Laboratory of Neuromuscular and Cardiovascular Study of Motion (LANECASM), Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis plan, and clinical study report may be shared when results will be published in a Journal.

REFERENCES:
- [Derived] Elpidoforou M, Grimani I, Papadopoulou M, Papagiannakis N, Bougea A, Simitsi AM, Sfikas E, Alexandratou I, Alefanti I, Antonelou R, Koros C, Mavroyianni I, Chrysovitsanou C, Stefanis L, Bakalidou D. An In-Person and Online Intervention for Parkinson Disease (UPGRADE-PD): Protocol for a Patient-Centered and Culturally Tailored 3-Arm Crossover Trial. JMIR Res Protoc. 2025 May 2;14:e65490. doi: 10.2196/65490. PMID 40314994